CLINICAL TRIAL: NCT04276597
Title: A Phase II, Non-Randomized, Open-Label, Single-center, Physician Sponsored Study to Determine the Safety and Effectiveness of Lu-177 DOTATOC in Adult Subjects With Somatostatin Receptor Expressing Pulmonary, Pheochromocytoma, paragangliomUnknown Primary, and Thymus Neuroendocrine Tumors (PUTNET) or Any Other Non-.GEP-NET.
Brief Title: Phase-II Study of Lu177DOTATOC in Adults With STTR(+)Pulmonary, Pheochromocytoma, Paraganglioma, Unknown Primary, Thymus NETs (PUTNET), or Any Other Non-.GEP-NET.
Acronym: PUTNET
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No subjects were eligible for the study. The study closed on 07-15-2021.
Sponsor: Excel Diagnostics and Nuclear Oncology Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 143631
Record Dates: First submitted 2020-02-14; First posted 2020-02-19 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Pulmonary Neuroendocrine Neoplasm; Pheochromocytoma; Paraganglioma; Thymus Carcinoid; Unknown Primary Tumors; Neuroendocrine Tumors; Neuroendocrine Skin Carcinoma; Neuroendocrine Breast Tumor; Neuroendocrine Carcinoma Metastatic; Neuroendocrine Neoplasm of Ovary
Keywords: Neuroendocrine tumors; Thymus neuroendocrine; Unknown Primary; Paraganglioma; Pheochromocytoma; Pulmonary; Any other non-.GEP-NET; NET
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma; Neoplasms, Unknown Primary; Neuroendocrine Tumors; Carcinoma, Merkel Cell | interventions — 177Lu-octreotide, DOTA(0)-Tyr(3)-

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lu177 DOTATOC treatment (Experimental): 4 doses of 200mCi 177Lu- DOTATOC PRRT
  Interventions: Drug: 177Lu-DOTATOC

INTERVENTIONS:
Drug: 177Lu-DOTATOC — 177Lu labeled somatostatin receptors targeting ligand

SUMMARY:
Determine the safety and effectiveness of Lu-177 DOTATOC in adult subjects with somatostatin receptor-expressing Pulmonary, Pheochromocytoma, Paraganglioma, Unknown primary, and Thymus neuroendocrine tumors or any other non-.GEP-NET.

The treatment regimen will consist of 4 doses of 200 (±10%) mCi 177Lu-DOTATOC administered at 8+/- 1-week intervals.

ELIGIBILITY:
Inclusion criteria:

* Signed informed consent.
* Subjects of either sex, aged ≥18 years.
* ECOG status 0-2.
* Life-expectancy of at least 12 weeks.
* Histologically/cytologically confirmed diagnosis of SSTR (+) neuroendocrine tumors of the lung, Pheochromocytoma, Paraganglioma, thymus, and unknown primary, unresectable or metastatic.
* Measurable disease per RECIST 1.1, on CT/MRI scans, defined as at least 1 lesion with ≥ 1 cm in longest diameter (lymph nodes along short axis >15 mm).
* Appropriate diagnostic imaging studies, at the discretion of the P.I. including but not limited to CT, MRI , 18F-FDG PET/CT, NAF PET/CT bone scan, ultrasound, etc. of the tumor region or suspected area within the 4 weeks of dosing day.
* Somatostatin receptor positive (SSTR+) disease, as evidenced by available FDA, commercially of IND approved SSTR imaging (SRI), within 4 weeks prior to the first cycle
* Recent blood test results (within 2weeks pre-dose) as follows:
* Sufficient bone marrow capacity as defined by WBC ≥2,500/µl and WBC≥2,000/mm3 for subsequent cycles; platelets ≥ 100,000 (100 * 103/mm3) for the first treatment and ≥75,000 for the subsequent therapies, Hgb ≥8.9 g/dl for the first treatment and 8.0 g/dl for the subsequent therapies, ANC ≥1500/mm3 for the first treatment and ≥1000/ mm3; for the subsequent therapies.
* ALT, AST values ≤3 times ULN
* Bilirubin: ≤3 times ULN
* Serum creatinine ≤ 150 µmol/liter or 1.7 mg/dl
* Negative pregnancy test in women capable of child-bearing within 48 hours of IMP administration.
* Serum albumin > 3.0g/L (<3 g/L may be acceptable at the discretion of investigator, if PT, PTT, and INR are within normal range)
* All available FDA-approved therapies for which the subject is eligible have been exhausted (with the exception of PRRT), unless available therapies are refused by the subject (with the exception of somatostatin analogue, octreotide, and somatuline).

Exclusion Criteria:

* Known hypersensitivity to any of the excipients of Lu-177 DOTATOC.
* Therapeutic use of any somatostatin analogue, including Sandostatin® LAR (within 28 days) and Sandostatin® (within 1 day) prior to treatment.
* Subjects with unusual hematological parameters, including an increased MCV (>105fL), and especially in those who had previous chemotherapy, the advice of a hematologist should be sought for adequate further work-up
* Any subject who is taking concomitant medications that decrease renal function (such as aminoglycoside antibiotics).
* Female subjects who are pregnant, lactating or women of childbearing potential not willing to practice effective contraceptive techniques during the study period and for 67 days (more than 10 half-lives of 177Lu after the last treatment, or male subjects who have female partners of childbearing potential not willing to practice abstinence or effective contraception, during the study period and for 67 days after the last treatment.
* Current somatic or psychiatric disease/condition that may interfere with the objectives and assessments of the study.
* Indication for surgical lesion removal with curative potential
* Planned (for the period of study participation): chemotherapy, immunotherapy, radiation therapy (unless regional for pain relief) chemo-embolization, bland embolization, radio-embolization, treatment with cyclosporine-A.
* Known brain metastases; unless these metastases have been treated and stabilized 6 months prior to enrolment
* Completion of: (1) cytotoxic chemotherapy for less than 6 weeks; (2) a biological agent for less than 5 half-lives; and (3) radiation therapy (except regional for pain relief) for less than 6 weeks prior to study enrolment,
* Uncontrolled congestive heart failure; subjects suspected of having this condition need to show ejection fraction of > 35% as determined by MUGA scan.
* Glomerular Filtration Rate (GFR) < 35 mL/min
* Subjects with prior peptide receptor radionuclide therapy (PPRT).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Assessment of the overall response rate | 12 monts
  determined using standard of care scans NETSPOT PET/CT, Octreoscan SPECT/CT, MRI

SECONDARY OUTCOMES:
Progression Free Survival (rPFS) in subjects receiving 4 cycles of therapy Monitoring of the changes in quality of life (QOL) through assessment of ECOG performance status and a QOL subject questionnaire. | 12 months
  determined using standard of care scans NETSPOT PET/CT, Octreoscan SPECT/CT, MRI

CONTACTS AND LOCATIONS:
Overall Officials: Ebrahim Delpassand, MD, Principal Investigator — Excel Diagnostics and Nuclear Oncology Center; Rodolfo Nunez, MD, Study Director — Excel Diagnostics and Nuclear Oncology Center; Afshin Shafie, MD, Study Director — Excel Diagnostics and Nuclear Oncology Center; Ayman Gaber, MD, Study Director — Excel Diagnostics and Nuclear Oncology Center
Locations (1):
- Excel Diagnostics and Nuclear Oncology Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No